CLINICAL TRIAL: NCT01186367
Title: Exercise Intensity Trial (EXCITE): A Randomized Trial Comparing the Effects of Linear Versus Nonlinear Aerobic Training in Women With Operable Breast Cancer
Brief Title: Trial Comparing the Effects of Linear Versus Nonlinear Aerobic Training in Women With Operable Breast Cancer
Acronym: Excite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-147
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; Linear Versus Nonlinear Aerobic Training; 15-147
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise Test; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Linear Aerobic Training (Experimental): The ultimate goal is for participants to complete approximately 130-180 minutes/week of aerobic training, at 60% to 75 % of the individually determined exercise capacity (VO2peak), for 16 weeks. VO2peak will be determined by the second CPET performed at baseline.
  Interventions: Behavioral: Linear Aerobic Training; Other: Cardiopulmonary exercise test (CPET); Other: Blood draws
- Nonlinear Aerobic Training (Experimental): The ultimate goal is for participants to complete approximately 130-180 minutes/week of aerobic training at 55% to 100% of the individually determined exercise capacity (VO2peak), for 16 weeks. VO2peak will be determined by the second CPET performed at Baseline and as well as the CPET performed at Midpoint.
  Interventions: Behavioral: Nonlinear Aerobic Training; Other: Cardiopulmonary exercise test (CPET); Other: Blood draws
- Progressive Stretching Group (Attention control) (Experimental): The ultimate goal for the progressive stretching program is 3 to 4 individual stretching sessions/week for 10 to 50 minutes per session (+/- 10 minutes).
  Interventions: Behavioral: Progressive Stretching; Other: Cardiopulmonary exercise test (CPET); Other: Blood draws

INTERVENTIONS:
Behavioral: Linear Aerobic Training — The 130-180 minutes/week will be achieved via either 3 to 4 individual aerobic training sessions at approximately 10 to 50 minutes per/session (± 10 minutes).
  Arms: Linear Aerobic Training
Behavioral: Nonlinear Aerobic Training — The 130-180 minutes/week will be achieved via 3 to 4 individual aerobic training sessions at approximately 10 to 50 minutes/ per session (+/- 10 minutes).
  Arms: Nonlinear Aerobic Training
Behavioral: Progressive Stretching — All sessions are required to be supervised. Duration of the stretching sessions is prescribed and implemented in accordance with standard stretching and flexibility training principles. This approach will be applied to guide each participant's prescribed stretching plan, with dose and scheduling modifications made by exercise physiologists, as required.
  Arms: Progressive Stretching Group (Attention control)
Other: Cardiopulmonary exercise test (CPET)
Other: Blood draws — Complete blood count

SUMMARY:
The purpose of this study is to compare the effects of 3 different approaches to exercise training in women with early stage breast cancer who have completed all primary treatments (except hormone therapy, if appropriate). Prior research in women with early stage breast cancer has shown that some treatments may have an adverse impact on physical fitness levels leading to feelings of fatigue and poor quality of life. Supervised exercise training has been shown to reduce some of these side-effects. However, all the exercise programs have followed essentially the same approach. This study is designed to see if a different approach to exercise training is more effective than the conventional approach currently in use.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45-80 years
* Female
* Has been diagnosed with early-stage breast cancer
* Post-menopausal, defined as :
* Age ≥ 45 with no menses for at least 2 years
* Chemically induced menopause through ovarian suppression, as determined by the primary oncologist
* An interval of at least one year, but no more than five years, following the full completion of primary therapy for malignant disease. Primary therapy is defined as:

  * Surgery plus radiation
  * Surgery plus chemotherapy
  * Surgery plus trastuzumab
  * Surgery plus hormone therapy Note: For patients who receive hormone therapy following surgery, the definition of one-year post-completion of therapy is defined by the surgery date. Patients who are currently receiving hormone therapy are eligible for enrollment.
* Weight of < 205 kgs
* ECOG status of 0 or 1
* Life expectancy ≥ 6 months
* Performing less than 150 minutes of structured moderate-intensity or strenuous intensity exercise per week.
* Exercise intolerance defined by a VO2peak below that predicted for sedentary age and sex-matched individuals as defined in Appendix H.
* Willing to be randomized to one of the study arms
* Able to complete an acceptable baseline CPET, in the absence of high risk ECG findings or other inappropriate response to exercise as determined by the investigator.
* Able to achieve an acceptable peak baseline CPET, as defined by any of the following criteria:

  * Achieving a plateau in oxygen consumption, concurrent with an increase in power output;
  * A respiratory exchange ratio ≥ 1.10;
  * Attainment of maximal predicted heart rate (HRmax) (i.e., within 10 bpm of age-predicted HRmax [HRmax = 220-Age[years]);
  * Volitional exhaustion, as measured by a rating of perceived exertion (RPE) ≥ 18 on the BORG scale.

Exclusion Criteria:

* Any of the following absolute contraindications to cardiopulmonary exercise testing:

  * Acute myocardial infarction within 3-5 days of any planned study procedures;
  * Unstable angina;
  * Uncontrolled arrhythmia causing symptoms or hemodynamic compromise;
  * Recurrent syncope;
  * Active endocarditis;
  * Acute myocarditis or pericarditis;
  * Symptomatic severe aortic stenosis;
  * Uncontrolled heart failure;
  * Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures
  * Thrombosis of lower extremities;
  * Suspected dissecting aneurysm;
  * Uncontrolled asthma;
  * Pulmonary edema;
  * Respiratory failure;
  * Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis);
* Presence of any other concurrent, actively treated malignancy
* History of any other malignancy treated within the past 3 years (other than non-melanoma skin cancer)
* Presence of metastatic disease
* Room air desaturation at rest ≤ 85%
* Mental impairment leading to inability to cooperate
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the participant a poor candidate for the trial

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-11-11 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Scott JM, Thomas SM, Peppercorn JM, Herndon JE 2nd, Douglas PS, Khouri MG, Dang CT, Yu AF, Catalina D, Ciolino C, Capaci C, Michalski MG, Eves ND, Jones LW. Effects of Exercise Therapy Dosing Schedule on Impaired Cardiorespiratory Fitness in Patients With Primary Breast Cancer: A Randomized Controlled Trial. Circulation. 2020 Feb 18;141(7):560-570. doi: 10.1161/CIRCULATIONAHA.119.043483. Epub 2020 Feb 17. PMID 32065769
- [Derived] Michalski M, Rowed K, Lavery JA, Moskowitz CS, Capaci C, Stene G, Edvardsen E, Eves ND, Jones LW, Scott JM. Validity of Estimated Cardiorespiratory Fitness in Patients With Primary Breast Cancer. JACC CardioOncol. 2022 Jun 21;4(2):210-219. doi: 10.1016/j.jaccao.2022.05.003. eCollection 2022 Jun. PMID 35818548
- [Derived] Jones LW, Douglas PS, Eves ND, Marcom PK, Kraus WE, Herndon JE 2nd, Inman BA, Allen JD, Peppercorn J. Rationale and design of the Exercise Intensity Trial (EXCITE): A randomized trial comparing the effects of moderate versus moderate to high-intensity aerobic training in women with operable breast cancer. BMC Cancer. 2010 Oct 6;10:531. doi: 10.1186/1471-2407-10-531. PMID 20925920
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Linear Aerobic Training: The ultimate goal is for participants to complete approximately 130-180 minutes/week of aerobic training, at 60% to 75 % of the individually determined exercise capacity (VO2peak), for 16 weeks. VO2peak will be determined by the second CPET performed at baseline.
  Linear Aerobic Training: The 130-180 minutes/week will be achieved via either 3 to 4 individual aerobic training sessions at approximately 10 to 50 minutes per/session (± 10 minutes).
  Cardiopulmonary exercise test (CPET)
  Blood draws: Complete blood count
- Nonlinear Aerobic Training: The ultimate goal is for participants to complete approximately 130-180 minutes/week of aerobic training at 55% to 100% of the individually determined exercise capacity (VO2peak), for 16 weeks. VO2peak will be determined by the second CPET performed at Baseline and as well as the CPET performed at Midpoint.
  Nonlinear Aerobic Training: The 130-180 minutes/week will be achieved via 3 to 4 individual aerobic training sessions at approximately 10 to 50 minutes/ per session (+/- 10 minutes).
  Cardiopulmonary exercise test (CPET)
  Blood draws: Complete blood count
- Progressive Stretching Group (Attention Control): The ultimate goal for the progressive stretching program is 3 to 4 individual stretching sessions/week for 10 to 50 minutes per session (+/- 10 minutes).
  Progressive Stretching: All sessions are required to be supervised. Duration of the stretching sessions is prescribed and implemented in accordance with standard stretching and flexibility training principles. This approach will be applied to guide each participant's prescribed stretching plan, with dose and scheduling modifications made by exercise physiologists, as required.
  Cardiopulmonary exercise test (CPET)
  Blood draws: Complete blood count
Period: Overall Study
Arm/Group | Linear Aerobic Training | Nonlinear Aerobic Training | Progressive Stretching Group (Attention Control)
Started | 58 | 59 | 57
Completed | 51 | 54 | 50
Not Completed | 7 | 5 | 7
Not completed — Lost to Follow-up | 7 | 4 | 7
Not completed — Did not receive study treatment | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Linear Aerobic Training | Nonlinear Aerobic Training | Progressive Stretching Group (Attention Control) | Total
Number analyzed (Participants) | 58 | 59 | 57 | 174
Age, Continuous [Mean (Full Range); unit: years] | 59 [44 to 76] | 58 [33 to 78] | 58 [38 to 73] | 58 [33 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 57 | 174
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 5
  Not Hispanic or Latino | 51 | 50 | 48 | 149
  Unknown or Not Reported | 6 | 6 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 10 | 12 | 35
  White | 38 | 40 | 37 | 115
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 6 | 6 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58 | 59 | 57 | 174

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Effect of High-intensity to Moderate-intensity Aerobic Training, Relative to Attention-control, on Peak Oxygen Consumption.
Description: VO2 or peak oxygen consumption will be measured at Baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Linear Aerobic Training | Nonlinear Aerobic Training | Progressive Stretching Group (Attention Control)
Number analyzed (Participants) | 58 | 59 | 57
mL/kg/min | 21.5 (4.4) | 22.2 (4.3) | 21.8 (3.8)

2. Primary Outcome: To Compare the Effect of High-intensity to Moderate-intensity Aerobic Training, Relative to Attention-control, on Peak Oxygen Consumption.
Description: VO2 or peak oxygen consumption for nonlinear aerobic training will be measured at mid-point (8 weeks)
Time Frame: 8 weeks
Population: Only nonlinear aerobic training measured at 8 weeks
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Linear Aerobic Training | Nonlinear Aerobic Training | Progressive Stretching Group (Attention Control)
Number analyzed (Participants) | 0 | 58 | 0
mL/kg/min |  | 22.6 (4.5) |

3. Primary Outcome: To Compare the Effect of High-intensity to Moderate-intensity Aerobic Training, Relative to Attention-control, on Peak Oxygen Consumption.
Description: VO2 or peak oxygen consumption will be measured at post-intervention (16 weeks).
Time Frame: 16 weeks
Population: Nonlinear aerobic training measured at 16 weeks
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Linear Aerobic Training | Nonlinear Aerobic Training | Progressive Stretching Group (Attention Control)
Number analyzed (Participants) | 58 | 59 | 57
mL/kg/min | 22.2 (4.6) | 23.1 (4.8) | 21.8 (3.7)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Linear Aerobic Training | Nonlinear Aerobic Training | Progressive Stretching Group (Attention Control)
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/59 | 1/57
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/59 | 0/57
Other Adverse Events (participants affected / at risk) | 58/58 | 59/59 | 8/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linear Aerobic Training (N=58) | Nonlinear Aerobic Training (N=59) | Progressive Stretching Group (Attention Control) (N=57)
Abnormal heart response (Cardiac disorders) | 5 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 15 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 2
Dizziness (Nervous system disorders) | 6 | 7 | 0
General fatigue (General disorders) | 7 | 7 | 1
Lower extremity fatigue (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Pain in extremity (Metabolism and nutrition disorders) | 14 | 10 | 2
Abnormal blood pressure response (Vascular disorders) | 1 | 1 | 1
Low oxygen saturation (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0 | 0
Other (General disorders) | 8 | 11 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT01186367/Prot_SAP_000.pdf